CLINICAL TRIAL: NCT01805973
Title: Surviving Aneurysm Surgery: A Pilot Randomised Controlled Trial on Exercise Training in Abdominal Aortic Aneurysm Patients
Brief Title: Surviving Aneurysm Surgery: A Pilot Study on Exercise Training in Abdominal Aortic Aneurysm Patients
Acronym: SAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013VSAS001
Record Dates: First submitted 2013-02-28; First posted 2013-03-06 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Aortic Aneurysm; Aortic Disease; Vascular Disease; Cardiovascular Disease
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Diseases; Vascular Diseases; Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Standard pre-operative care, no active intervention
- Exercise Training (Experimental): Supervised Exercise Training Programme Patients will be required to attend three 50 minute exercise sessions per week for 18 weeks. They will exercise in groups of 8-12 and will be supervised by an experienced exercise physiologist. Each session will comprise a 15 minute warm up, 30 minutes of moderate intensity aerobic exercise followed by a 10 minute cool down period.
  The patients will have the option to choose from three different exercise programmes tailored to individuals of mixed abilities (and co-morbidities).
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training — Patients will participate in a supervised exercise training programme for 18 weeks. Patients will participate in a 50 minute exercise regime three times a week.
  Arms: Exercise Training

SUMMARY:
An abdominal aortic aneurysm (AAA) is an enlargement or ballooning of the main artery supplying high pressure blood from the heart to the body. AAAs may continue to stretch until they burst (rupture) causing 7000 deaths per year in the United Kingdom (UK); 2.1% of all deaths in men over 65. Planned repair before rupture is critical and the National AAA Screening Programme (NAAASP) is being introduced to identify AAAs in men before rupture. Screening will identify over 9000 men per year with a previously undiagnosed AAA. More than 90% of screen detected AAAs are small, do no require repair, enter ultrasound follow-up (surveillance) and may benefit from exercise to improve fitness before repair.

Over 4000 elective AAA repairs per year are performed in the UK and it has been suggested that exercise training and weight loss may reduce mortality and complications of AAA repair. This pilot study will examine the feasibility of supervised exercise training for patients with AAAs and determine the optimal duration of training to achieve worthwhile improvements in fitness.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) affects 4% of men aged 65-79, a prevalence rising as our population ages. As most patients suffering rupture die immediately, elective AAA repair is critical and the National AAA Screening Programme (NAAASP) is being implemented across the UK to identify AAAs for elective repair. Manchester is the first major urban population to be screened. The UK had the highest mortality rates following elective open AAA repair in Europe (7% v 3.5%); the AAA Quality Improvement Programme's (AAAQIP) target is to reduce this to under 3.5% by 2013.

The benefits of exercise across a broad spectrum of medical conditions are now increasingly recognised; especially in the elderly. Exercise training may reduce mortality and complications in major surgery. Cardiopulmonary exercise testing (CPET) measures cardiopulmonary reserve and predicts outcome in major surgery. The Manchester CPET study group demonstrated that anaerobic threshold (AT) and peak oxygen consumption (VO2 peak) predict 30 and 90-day mortality in elective AAA repair.

The investigators propose a pilot randomised controlled trial (RCT) to determine whether a structured exercise programme improves fitness measured by CPET, and the optimal duration of training for AAA surgery. As over 90% of AAAs detected by screening are < 5.5cm and enter surveillance, these patients offer a unique opportunity to explore the ideal duration of exercise training as surgery is not indicated for months or years.

100 participants on AAA surveillance will be recruited and randomised to either exercise training or standard preoperative care (50 in each arm) to answer the following research questions:

1. Can a supervised exercise programme improve performance in CPET measures that predict outcome in AAA surgery?
2. What is the optimal period of training needed to achieve a significant improvement in CPET scores?
3. How long is any exercise-induced improvement in fitness sustained?
4. The economic and health costs of a supervised exercise training programme

Exercise subjects will attend a 60 minute supervised exercise programme of moderate intensity (70% of heart rate reserve) x3/week at a local gym. All participants will undergo CPET assessment of cardiopulmonary fitness and complete a health-related quality of life (Medical Outcomes Study 36-Item Short-Form Health Survey) at baseline and 18 weeks. The exercise subjects will undergo further CPET studies at 6, 12 and 36 weeks to investigate the duration of training needed to optimise fitness and the length of time improvements in fitness persist. Other important health related outcomes include blood pressure and lipid profile and frequency of health service visits (e.g. General Practitioner appointments) will be recorded for all participants at baseline and 18 weeks to provide data on the effects of exercise on health care costs. Longitudinal regression models, with Normal and Poisson distributions as appropriate, will be used to assess differences between the groups with respect to CPET changes, other health-related outcomes and frequency of health service visits over the whole study period. This pilot study will also explore strategies to encourage participation and compliance with exercise which may also improve general health outcomes and save National Health Service (NHS) costs by reducing demand.

The overall aim is to collect the data needed to design a definitive multicentre trial on whether physical exercise reduces morbidity and/or mortality in AAA repair.

Those aged >65 are the fastest growing segment of our population. This pilot study will contribute to public health policy drive on the impact of physical activity on functional capacity, quality of life and independence.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with an AAA ≥3.5cm to <5.5cm in men and ≥3.5cm to <5.0cm in women
* Age 50-85 years and willing to consider exercise training
* Fit for either open or Endovascular Aneurysm Repair AAA repair

Exclusion Criteria:

* Unable to participate in an exercise test or inability to exercise consistently because of musculoskeletal or other health problems
* History of severe liver disease (INR>2, serum albumin <3.0g/dL, jaundice)
* Unstable angina: Patients with angina of less than 2 months' duration, severe or occurring three or more times per day, or angina that is becoming either more frequent of precipitated by less exertion or angina at rest
* Uncontrolled atrial fibrillation (AF) or other arrhythmia: Untreated episodes of paroxysmal AF in the last 3 months
* Moderate or severe aortic valve stenosis (peak systolic pressure gradient > 40mmHg and with an aortic valve area of <1cm^2.
* Class III/IV heart failure and / or an ejection fraction <25%
* Active pericarditis or myocarditis
* CPET induced ischaemia
* Diagnosis or treatment for a malignancy (excluding skin) over the previous 12 months

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test Score | 18 weeks
  The investigators will determine if supervised exercise training improves cardiopulmonary fitness. Peak oxygen uptake and ventilatory threshold will be assessed during an incremental-load cycling test.

SECONDARY OUTCOMES:
Cardiopulmonary Exercise Test Score | 12 weeks
  For the intervention (exercise) arm the investigators will assess the CPET score at 6 and 12 weeks to determine the optimal duration of exercise training.
  Peak oxygen uptake and ventilatory threshold will be assessed during an incremental-load cycling test.
Cardiopulmonary Exercise Test Score | 36 weeks
  The investigators will determine how long any improvements in fitness are sustained after exercise is stopped.
  Peak oxygen uptake and ventilatory threshold will be assessed during an incremental-load cycling test.
Health-related quality of life | 18 weeks
  Fasting blood samples will be taken to assess changes in lipid profile and other biomarkers of cardiovascular disease.
  Blood pressure control will be monitored.
Quality of Life | 18 weeks
  Health-related quality of life will be assessed using the Medical Outcomes Study Short Form-36 questionnaire.
Cost | 18 weeks
  A preliminary economic analysis will be performed to determine the cost of prescribed exercise training before surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Charles M McCollum, MD, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- University Hospital of South Manchester NHS Foundation Trust, Manchester, Lancashire, United Kingdom